CLINICAL TRIAL: NCT07011745
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of KarXT + KarX-EC for the Treatment of Agitation Associated With Alzheimer's Disease
Brief Title: A Phase 3 Study to Evaluate the Safety and Efficacy of KarXT + KarX-EC for the Treatment of Agitation Associated With Alzheimer's Disease (ADAGIO-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0024; 2025-520613-31 (Other: EU CTR); U1111-1316-5745 (Other: WHO)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT + KarX-EC (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride Capsule; Drug: Xanomeline Enteric Capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xanomeline/Trospium Chloride Capsule — Specified dose on specified days
  Other Names: KarXT; BMS-986510
  Arms: KarXT + KarX-EC
Drug: Xanomeline Enteric Capsule — Specified dose on specified days
  Other Names: KarX-EC; BMS-986519
  Arms: KarXT + KarX-EC
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KarXT + KarX-EC in adult participants with agitation related to Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria

- A diagnosis of Alzheimer's disease (AD) in accordance with the 2024 Alzheimer's Association criteria with one of the following confirmations of AD pathology:

i) Historical evidence of AD diagnosis with amyloid positron emission tomography (PET), Aβ42/40 ratio in CSF, pTau181/Aβ42 ratio in CSF or pTau217/Aβ42 ratio in plasma using an Health Authority (HA)-authorized diagnostic assay.

ii) If no historical evidence available:

A. A plasma biomarker will be assessed for eligibility if allowed per regulatory requirements. The test cutoff(s) will be based on diagnostic use approval.

B. If a plasma biomarker assay cannot be used or if the assay result is inconclusive, conduct one the following:

* Amyloid PET.
* Aβ42/40 ratio or pTau181/Aβ42 ratio in CSF using an HA-authorized diagnostic assay.

  * Mini-Mental State Examination (MMSE) score of 5 to 22, inclusive, at Screening (Visit 1).
  * Have one identified caregiver who should have sufficient contact (approximately 10 hours a week or more) and is willing to:

    i) Attend all visits and report on participant's status.

ii) Oversee participant compliance with medication and study procedures.

iii) Participate in the study assessments and provide informed consent to participate in the study.

* History of agitation that meets the International Psychogeriatric Association (IPA) consensus definition for agitation in cognitive disorders with onset at least two weeks prior to Screening (Visit 1).
* AD participants are required to have NPI/NPI-NH Agitation/Aggression score ≥ 4 at Screening (Visit 1) and Baseline (Visit 2).
* CGI-S ≥ 4, as related to agitation, at Screening (Visit 1) and Baseline (Visit 2).
* At least 1 of the following 3 criteria must be established from the CMAI-IPA at Screening (Visit 1) and Baseline (Visit 2; CMAI-IPA Physical/Verbal Aggression Positivity):

  i) 1 or more aggressive behaviors occurring at least several times per week.

ii) 2 or more aggressive behaviors occurring at least once or twice per week.

iii) 3 or more aggressive behaviors occurring less than once per week.

Exclusion Criteria

- Medical Conditions.

i) Agitation symptoms that are primarily attributable to a condition other than the AD causing the dementia.

ii) History of bipolar disorder, schizophrenia, or schizoaffective disorder.

iii) History of (or at high risk for) urinary retention, gastric retention, or narrow-angle glaucoma as evaluated by the Investigator.

iv) Risk of suicidal behavior during the study as determined by the Investigator's clinical assessment and/or C-SSR.

- Prior/Concomitant Therapy.

i) Recent history of receiving monoamine oxidase inhibitors, anticonvulsants (eg, lamotrigine, divalproex), mood stabilizers (eg, lithium), tricyclic antidepressants (eg, imipramine, desipramine), or any other psychoactive medications except for as needed anxiolytics (eg, lorazepam).

A. Selective serotonin reuptake inhibitors and serotonin norepinephrine reuptake inhibitors taken at a stable dose for at least 8 weeks prior to Screening (Visit 1) may be permitted.

B. Mirtazapine or trazodone may be used as a hypnotic if started at least 8 weeks prior to Screening (Visit 1).

- Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2028-11-03 (Estimated); Study Completion 2028-11-13 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the Cohen-Mansfield Agitation Inventory-International Psychogeriatric Association (CMAI-IPA) total score at Week 14 | At Week 14

SECONDARY OUTCOMES:
Change from baseline on the Clinical Global Impressions-Severity (CGI-S) at Week 14 | At Week 14
Change from baseline on CMAI-IPA Domains at Week 14 | At Week 14
Change from baseline on CMAI Total Score at Week 14 | At Week 14
Number of participants with Occurrence of Response at Week 14 | At Week 14
  As determined by CMAI-IPA changes of at least 30%, 40%, and 50% from baseline
Change from baseline on the Neuropsychiatric Inventory/Neuropsychiatric Inventory -Nursing Home (NPI/NPI-NH) Total Score at Week 14 | At Week 14
Number of participants with Adverse Events (AEs) | Up to Week 18
Number of participants with Treatment Emergent AEs (TEAEs) | Up to Week 18
Number of participants with Serious AEs (SAEs) | Up to Week 18
Number of participants with AEs leading to study drug withdrawal | Up to Week 18
Number of deaths | Up to Week 18
Number of participants with AEs of Special Interest (AESIs) | Up to Week 18
Barnes Akathisia Rating Scale (BARS) | Up to Week 18
Abnormal Involuntary Movement Scale (AIMS) | Up to Week 18
Body weight | Up to Week 18
Body Mass Index (BMI) | Up to Week 18
Number of participants with vital sign abnormalities | Up to Week 18
Number of participants with clinical laboratory abnormalities | Up to Week 18
Number of participants with electrocardiogram (ECG) abnormalities | Up to Week 18
Number of participants with suicidal ideation as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Week 18
Severity of benign prostatic hyperplasia in male participants as assessed by International Prostate Symptom Score (IPSS) | Up to Week 18

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (139):
- United States (37):
  - Chandler Clinical Trials, LLC, Chandler, Arizona
  - Local Institution - 2631, Chandler, Arizona
  - Local Institution - 2625, Long Beach, California
  - Local Institution - 2607, Long Beach, California
  - Local Institution - 2642, Long Beach, California
  - Local Institution - 2627, Napa, California
  - Local Institution - 2613, Pasadena, California
  - Local Institution - 2614, San Diego, California
  - Alliance Clinical -West Hills, West Hills, California
  - Local Institution - 2601, Basalt, Colorado
  - Local Institution - 2635, Colorado Springs, Colorado
  - Local Institution - 2632, Norwalk, Connecticut
  - Envision Trials LLC, Bonita Springs, Florida
  - Key Clinical Research, Bradenton, Florida
  - Local Institution - 2636, Doral, Florida
  - Local Institution - 2606, Homestead, Florida
  - Local Institution - 2633, Miami, Florida
  - Local Institution - 2637, Miami, Florida
  - Local Institution - 2634, Orlando, Florida
  - IPTB Clinical Research, Tampa, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Vitalix Clinical, Worcester, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Local Institution - 2630, Saint Paul, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Sharlin Health Neuroscience Research Center, Ozark, Missouri
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - Richmond Behavioral Associates, Staten Island, New York
  - West Clinical Research, Morehead City, North Carolina
  - Velocity Clinical Research - Blue Ash, Blue Ash, Ohio
  - Epic Medical Research, LLC - Carrolton, Carrollton, Texas
  - Horizon Clinical Research Center - Houston, Cypress, Texas
  - Epic Medical Research, LLC - Mesquite, Mesquite, Texas
  - Local Institution - 2623, San Antonio, Texas
  - Pantheon Clinical Research, LLC, Bountiful, Utah
  - Local Institution - 2638, Kirkland, Washington
  - Local Institution - 2610, Milwaukee, Wisconsin
- Argentina (7):
  - Local Institution - 2005, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 2006, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 2004, Buenos Aires
  - Local Institution - 2000, Córdoba
  - Local Institution - 2002, Córdoba
  - Local Institution - 2003, Córdoba
  - Local Institution - 2001, Mendoza
- Chile (6):
  - Local Institution - 2055, Viña del Mar, Región de Valparaíso
  - Local Institution - 2051, Santiago, Santiago Metropolitan
  - Local Institution - 2050, Santiago, Santiago Metropolitan
  - Local Institution - 2052, Santiago, Santiago Metropolitan
  - Local Institution - 2054, Vitacura, Santiago Metropolitan
  - Local Institution - 2053, Antofagasta
- Czechia (9):
  - AGE Centrum, Olomouc, Olomoucký kraj
  - Neuropsychiatrie, Prague, Praha 6
  - Institut neuropsychiatricke pece (INEP), Praha, Prague, Praha 8
  - Neuro Health Centrum s.r.o., Brno, South Moravian
  - NEUROHK, Choceň
  - A-SHINE s.r.o., Pilsen
  - Local Institution - 2102, Prague
  - Local Institution - 2105, Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- France (7):
  - Centre Hospitalier Universitaire Toulouse - Cité de la Santé, Toulouse, Haute-Garonne
  - Local Institution - 2151, Villeurbanne, Rhône
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Roger Salengro, Lille
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren, Limoges
  - Local Institution - 2157, Montpellier
  - Local Institution - 2152, Paris
  - Les Hôpitaux Universitaires de Strasbourg - Hôpital de la Robertsau, Strasbourg
- Germany (4):
  - Local Institution - 2203, Erbach im Odenwald, Hesse
  - Local Institution - 2201, Düsseldorf
  - Local Institution - 2205, Halle
  - Local Institution - 2206, Westerstede
- Hungary (8):
  - Local Institution - 2257, Kalocsa, Bács-Kiskun county
  - Local Institution - 2250, Győr, Győr-Moson-Sopron
  - Local Institution - 2254, Gyöngyös, Heves County
  - Local Institution - 2256, Budapest
  - Local Institution - 2255, Budapest
  - Local Institution - 2251, Budapest
  - Local Institution - 2253, Budapest
  - Local Institution - 2252, Debrecen
- Israel (6):
  - The Chaim Sheba Medical Center, Ramat Gan, Central District
  - Local Institution - 2302, Petch Tikva, IL
  - Local Institution - 2301, Jerusalem
  - Sanz MC, Laniado Hospital, Netanya
  - The Israeli Alzheimer Medical Center, Ramat Gan
  - Bayit Balev Ltd., Rishon Le'Tzion
- Italy (8):
  - University of Naples Federico II, Napoli, Campania
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I - Viale del Policlinico 155, Rome, Lazio
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Rome, Lazio
  - Auxologico IRCCS - Auxologico San Luca, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, PI
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Local Institution - 2355, Isernia
  - Fondazione Policlinico Gemelli IRCCS, Roma
- Poland (7):
  - Centrum Medyczne HCP Szpital im. Jana Pawla II, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne NEUROMED, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - M2M Med, Chorzów
  - Centrum In Psyche Spersonalizowanej Psychiatrii I Terapii, Katowice
  - Local Institution - 2451, Lublin
  - Local Institution - 2452, Lublin
  - RCMed Oddzial Sochaczew, Sochaczew
- Puerto Rico (3):
  - Local Institution - 2641, San Juan
  - Local Institution - 2640, San Juan
  - Local Institution - 2639, San Juan
- South Korea (10):
  - Inha University Hospital, Incheon, Incheon Gwang'yeogsi
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Konkuk University Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 2406, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kyungpook National University Chilgok Hospital, Deagu, Taegu-Kwangyǒkshi
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - SMG-SNU Borame Medical Center, Seoul
  - The Catholic University of Korea, Yeouido St.Mary's Hospital, Seoul
- Ukraine (17):
  - Local Institution - 2555, Smila, Cherkasy Oblast
  - Local Institution - 2554, Dnipro, Dnipropetrovsk Oblast
  - Local Institution - 2561, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Local Institution - 2559, Skarzhyntsi, Khmelnytskyi Oblast
  - Local Institution - 2556, Hlevakha, Kyiv Oblast
  - Local Institution - 2566, Hlevakha, Kyiv Oblast
  - Local Institution - 2553, Kyiv, Kyivska Oblast
  - Local Institution - 2552, Lviv, Lviv Oblast
  - Local Institution - 2558, Lviv, Lviv Oblast
  - Local Institution - 2569, Lviv, Lviv Oblast
  - Local Institution - 2567, Oleksandrivka, Odesa Oblast
  - Local Institution - 2557, Poltava, Poltava Oblast
  - Local Institution - 2551, Vinnytsia, Vinnytsia Oblast
  - Local Institution - 2560, Lutsk, Volyn Oblast
  - Local Institution - 2550, Kropyvnytskyi
  - Local Institution - 2565, Kyiv
  - Local Institution - 2568, Odesa
- United Kingdom (10):
  - Local Institution - 2505, Preston, Lancashire
  - Surrey and Borders Partnership NHS Foundation Trust, Chertsey, Surrey
  - Local Institution - 2502, Cambridge
  - South London and Maudsley NHS Foundation Trust, London
  - Local Institution - 2500, London
  - NeuroClin Glasgow, Motherwell
  - Cornwall Partnership NHS Foundation Trust, Redruth
  - Sheffield Health and Social care NHS Foundation Trust, Sheffield
  - Local Institution - 2509, Stafford
  - Local Institution - 2503, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07011745.html